CLINICAL TRIAL: NCT03647800
Title: Phase 1B Open-Label, Dose-Escalation and Dose-Expansion Study of APVO436 in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) or High-Grade Myelodysplastic Syndrome (MDS)
Brief Title: Study of APVO436 in Patients With AML or MDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aptevo Research and Development LLC (Industry)
Responsible Party: Sponsor
Organization: Aptevo Therapeutics (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 5001
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: AML; MDS
Keywords: APVO436

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 parts. The first part of this Phase 1B study is an open-label, multiple dose ascending dose escalation phase to determine the recommended dose (RP2D) level of APVO436 for future Phase 2 studies. The goal of the dose expansion phase of the study (Part 2) is to (i) evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care and (ii) obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental monotherapy and combination therapy modalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PART 1 Dose Escalation - 10 dose cohorts (Experimental): CD123 and CD3 epsilon bispecific antibody
  Interventions: Biological: APVO436
- PART 2 Dose expansion - 5 cohorts (Experimental): 90 patients, 18/cohort in 5 dose expansion cohorts, will receive the recommended dose of APVO436 determined from Part 1
  Interventions: Biological: APVO436

INTERVENTIONS:
Biological: APVO436 — APVO436

SUMMARY:
The primary objective of the Phase 1 part of the study is to determine the recommended dose of APVO436 administered intravenously to patients with AML or MDS. The primary objective of the Phase 1b part of the study is to evaluate the clinical activity of APVO436 in patients with AML or MDS.

APVO436 is being studied in this Phase 1b, open-label, multi-center, two-part dose-escalation/dose expansion study to evaluate the safety, pharmacokinetic/pharmacodynamic (PK/PD), and clinical activity of APVO436 in patients with AML and MDS. The study will be conducted in 2 parts. The first part of this Phase 1B study is an open-label, multiple dose ascending dose escalation phase to determine the recommended dose (RP2D) level of APVO436 for future Phase 2 studies. The goal of the dose expansion phase of the study (Part 2) is to (i) evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care and (ii) obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental monotherapy and combination therapy modalities.

Study Objectives for Dose Escalation Phase

* Primary Objectives are to:

  1. Determine the RP2D level of APVO436 administered intravenously (IV) in patients with AML or MDS, and
  2. Evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care and obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental monotherapy and combination therapy modalities.
* Secondary Objectives are to:

  1. Define the safety profile and immunogenicity of APVO436; to determine the PK/PD of APVO436; to evaluate the clinical activity of APVO436 in AML and MDS patients.
  2. Further evaluate the safety profile and immunogenicity of APVO436 and the PK/PD of APVO436 and the relationship between PK/PD and clinical response.

Study Objectives for Dose Expansion Phase

* Primary Objective is to evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care.
* Secondary Objective is to obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental monotherapy and combination therapy modalities.

DETAILED DESCRIPTION:
Part 1 - Dose Escalation:

Dosing will start at the minimum anticipated biologic effect level (MABEL) in single-patient cohorts for the first 3 dose cohorts up to and including 3 mcg. Patients enrolled will have either: 1) relapsed or refractory AML and refuse or are not eligible for intensive chemotherapy or an allogeneic stem cell transplant, or 2) relapsed or refractory MDS and have > 5% blasts in the marrow or any circulating blasts in the peripheral blood and have failed a prior hypomethylating agent (HMA); failure is defined as intolerance to HMA, lack of response (no CR by at least 6 cycles), or have IWG defined progressive disease during or after treatment with an HMA.

In single-patient Cohorts 1 to 3, the next dose cohort will only enroll after the patient in the current dose cohort has completed the first cycle of dosing (4 weeks) and no Grade ≥ 2 adverse events (AEs) (hematologic or non-hematologic) have occurred. If any Grade ≥ 2 AE occurs in the single-patient cohorts, then that cohort and all subsequent single-patient cohorts will be expanded to a 3 + 3.

The next dose cohort in the 3 + 3 cohorts (all cohorts beyond Cohort 4) is started after patients in the previous dose cohort have completed the first cycle of dosing and an evaluation of AEs for DLTs during the DLT observation period has been completed. For the first 2 patients within each dose cohort, administration of the first dose must be separated by a minimum of 36 hours. At the conclusion of each cycle, patients with significant cytopenias without evidence of leukemia will have the dose delayed.

Beginning in Cohort 5, and for all cohorts going forward, stepped dosing will be introduced to mitigate against the development of infusion-related reactions and cytokine release syndrome.

Patients will receive APVO436 intravenously for six 28 day cycles, unless disease progression, intolerable toxicity, or withdrawal of consent occurs earlier. There is an option for longer treatment if the patient is responding. The RP2D level will be based on clinical activity, safety, incidence of DLTs, PK, and PD in each dose cohort.

Part 2 - Dose Expansion:

The MTD for APVO436 was not reached at a dose level of 240 µg/cycle (Cohort 10 in the dose escalation phase). The sub-MTD dose level of Cohort 6A was identified as the RP2D level of APVO436 for further evaluation during the expansion phase.

In the open-label, multi-center, dose expansion phase of the study (Part 2), a total of 90 primary AML patients will be enrolled into 5 cohorts of 18 patients each. The goal of this expansion phase of the study is to evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care and obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental monotherapy and combination therapy modalities.

In Cohorts 1-4, APVO436 will be administered at a fixed dosage of 18 mcg after a weekly ramp up during Cycle 1 (Cohorts 1, 3, 4) or Cycle 1-2 (Cohort 2). In Cohort 5, APVO436 will be administered at a fixed dose of 18 mcg twice weekly after a weekly ramp up during Cycle 1.

The specific patient populations and experimental treatments for the expansion phase are as follows:

Cohort 1. Induction with Chemotherapy (ChT) plus APVO436. 1st or 2nd Early Relapse. Patients may receive either Ara-C intermediate dose (IDAC) or MEC as the ChT backbone. Fit primary or secondary AML patients (Age: >18 years) in 1st or 2nd relapse with last CR <12 months or primary refractory disease will receive 4 x 28-day cycles of combined 2-drug immunochemotherapy: APA [APVO436+Intermediate dose ARA-C (IDAC) or APMEC [APVO436+MEC].

Cohort 2. Induction with APVO436 + Venetoclax + Azacitidine - Frontline or 1st Relapse. Poor prognostic but fit primary or secondary AML patients (Age >18 years) who are treatment-naïve or in 1st relapse will receive 4 x 28-day cycles of combined 3-drug immunochemotherapy: APVA [APVO436+Venetoclax+Azacitidine].

Cohort 3: Consolidation post 7+3 - Frontline + 1st Relapse. Fit primary AML patients (Age: >18 years) with FLT3-negative intermediate or adverse risk AML (including but not limited to: TP53, RUNX1 and ASXL1 mutations and/or complex cytogenetics) who are treatment-naïve or in 1st relapse with a duration of CR1<1 year will receive 4 x 28-day cycles of immunotherapy with APVO436 after hematologic recovery (ANC>1,000/µL; Hgb ≥9 g/dL; Plt≥100,000/µL) post induction.

Cohort 4: MRD-positive (MRD+) 1st Remission, APVO436 + Azacitidine combination. >18 years old MRD+ (at ≥0.1% level by multicolor-multiparameter flow cytometry [MFC] in Central Lab) high-risk 1st remission AML patients will be treated with 4 x 28-day cycles of APVO436 + oral azacitidine (Onureg, CC-486).

Cohort 5: MRD+ 2nd Remission, Single Agent APVO436. >18 years old MRD+ (at ≥0.1% level by MFC in Central Lab) AML patients who are in 2nd remission post-induction with a standard of care regimen will be treated with 4 x 28-day cycles of APVO436 monotherapy.

ELIGIBILITY:
Inclusion Criteria for Part 1: Dose Escalation Phase:

All patients must meet the following criteria prior to the first dose of study drug:

1. Signed informed consent. Consent must be obtained prior to any study-related procedure.
2. Age ≥ 18 years
3. Histologically confirmed AML or MDS:

   1. AML - relapsed or refractory AML and refuses or is not a candidate for intensive chemotherapy (due to prior failure or not eligible due to expected intolerance) or allogeneic transplant
   2. MDS - relapsed or refractory MDS with > 5% blasts in the marrow or any blasts in the peripheral blood. Patients must have failed prior treatment with an HMA (azacitidine, decitabine, or other HMA agent); failure is defined as intolerance to HMA, lack of response (no CR by at least 6 cycles), or have IWG-defined progressive disease during or after treatment with an HMA.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
5. Life expectancy of > 2 months in the Investigator's opinion
6. White blood cells (WBC) ≤ 25,000 cells/mm3 (may receive hydroxyurea to bring WBC count down prior to and during the first cycle of treatment with study drug if necessary)
7. Creatinine ≤ 2 × upper limit of normal (ULN)
8. Adequate liver test parameters: total bilirubin < 2.5 × ULN (if disease related or secondary to Gilbert's disease, then total bilirubin < 3.5 mg/dL), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) < 3 × ULN
9. Prothrombin time (PT) / international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 × ULN
10. Patients and partners of childbearing potential must be willing to use adequate contraception during the study and for 2 months after last study drug administration. Adequate contraception means less than 1% chance of pregnancy may occur with proper use of the method(s).

Exclusion Criteria for Part 1: Dose Escalation Phase:

A patient is not eligible to enroll into the study if they have any of the following:

1. Any CNS (cerebral/meningeal) disease related to underlying malignancy
2. History of seizures
3. Acute promyelocytic leukemia
4. Prior anti-CD123 therapy outside of this study
5. Any clinically significant graft-versus-host disease (GVHD) secondary to prior allogenic transplant. Patients must be > 90 days from transplant and have been on no immunosuppressive therapy for > 30 days. Topical corticosteroids for minor skin rash (<5% body surface area) is acceptable. Prior solid organ transplant is acceptable provided the patient is on no immunosuppressive therapy.
6. Any therapy or experimental treatment for MDS or AML within 7 days of the first dose of study drug. Must have recovered to Grade ≤ 1 from any Grade 2 to 4 toxicity from previous treatment. The use of hydroxyurea is acceptable and does not exclude the patient.
7. Active, uncontrolled infection requiring systemic therapy. If the infection is controlled or has resolved, maintenance and/or prophylactic systemic antimicrobials are permitted.
8. Major surgery within 3 weeks prior to first dose of study drug
9. Known to be positive for HIV, hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV)
10. Pregnant or breast feeding
11. Any other active systemic malignancies. Exceptions: noninvasive non-melanoma skin cancer, in situ carcinoma, cervical intraepithelial neoplasia, and breast or prostate cancer that is well controlled with anti-hormonal therapy
12. Any current autoimmune disorder requiring immunosuppressive therapy
13. Requires more than a replacement dose of corticosteroids (i.e., > 10 mg/day of prednisone or equivalent)
14. Any uncontrolled medical condition, including but not limited to:

    1. Symptomatic congestive heart failure ≥ Class III (New York Heart Association Functional Classification)
    2. Uncontrolled hypertension
    3. Unstable angina
    4. Myocardial infarction within previous 6 months
    5. Clinically significant arrhythmias not controlled by medication
    6. Uncontrolled metabolic disorders such as hypercalcemia
15. Substance use disorder, psychiatric, cognitive, or any other condition that, in the opinion of the Investigator, would pose a risk to the patient's safety, may compromise the patient's ability to understand and comply with the protocol or provide informed consent, or interfere with the study evaluation
16. Any difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration, or may cause a safety concern for the patient

Inclusion Criteria for Part 2: Dose Expansion Phase

Individuals eligible to participate in this study must meet all of the following:

All patients must meet the following criteria prior to the first dose of study drug:

1. Signed informed consent. Consent must be obtained prior to any study-related procedure.
2. Age: >18 years
3. Histologically confirmed AML: Subjects must have de novo (primary) AML (any WHO 2016 classification excluding acute promyelocytic leukemia, AML with myelodysplasia-related features, and Therapy-related secondary AML (except in Cohort 1 or Cohort 2)
4. Cohort 1: Fit primary or secondary AML patients (Age: >18 years) in 1st or 2nd relapse with last CR <1 year or primary refractory disease; Relapsed patients must have relapsed a maximum of two times after standard induction therapy for AML;
5. Cohort 2: Poor prognostic but fit primary or secondary AML patients who are treatment-naïve or in 1st relapse; patients in relapse must have relapsed only once after induction/consolidation therapy for AML, i.e., they must be in 1st relapse
6. Cohort 3: Fit primary AML patients with FLT3-negative intermediate or adverse risk AML (including but not limited to: TP53, RUNX1 and ASXL1 mutations and/or complex cytogenetics) who are treatment-naïve or in 1st relapse with a duration of CR1<1 year
7. Cohort 3: Patients are required to be either not in CR or be in CR is MRD positive (≥01% level) by MFC (Central Laboratory) post induction/consolidation to be eligible for APVO436 treatments.
8. Cohort 4: MRD+ (at ≥0.1% level by multicolor-multiparameter flow cytometry [MFC] in Central Lab) high-risk 1st remission AML patients
9. Cohort 4: Patients must be newly diagnosed AML patients in 1st remission who achieved their first remission after standard chemotherapy with a standard induction regimen with or without post-induction consolidation.
10. Cohort 5: Patients must be AML patients who were in 1st relapse and achieved a 2nd remission after standard chemotherapy with a standard induction regimen with or without post-induction consolidation.
11. Cohorts 1-5: If patient was treated with Cytarabine-containing induction or consolidation regimen, a minimum of 21 days must have passed since the last Cytarabine dose to allow for resolution of the side effects
12. Cohorts 1-3: Patients must have CD123-positive AML as confirmed by flow cytometry in Central Laboratory
13. Cohorts 4 and 5: Patients archived bone marrow or peripheral blood leukemic blast cells must be CD123-positive - local laboratory results are acceptable. If cells are available, the positivity should be confirmed by Central Laboratory.
14. Patients with precedent MDS are not eligible
15. MRD+ AML patients in Cohort 4 or Cohort 5 must be in CR (CR/CRi) for no more than 6 months and be MRD+, as determined by central hematopathology laboratory
16. MRD+ AML patients in Cohort 4 or Cohort 5 must first have an evaluable screening bone marrow sample confirmed as MRD+ by central hematopathology laboratory
17. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
18. Life expectancy of > 2 months in the Investigator's opinion
19. Creatinine ≤ 2 × upper limit of normal (ULN)
20. Adequate liver test parameters: total bilirubin < 2.5 × ULN (if disease related or secondary to Gilbert's disease, then total bilirubin < 3.5 mg/dL), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) < 3 × ULN
21. Prothrombin time (PT) / international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 × ULN
22. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) may participate, provided they meet the following conditions:

    1. Must agree to use physician-approved contraceptive methods (e.g., abstinence, intrauterine device, oral contraceptive, double barrier device) throughout the study and for 3 months following the last dose of APVO436; and
    2. Must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this study.
23. Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 3 months following the last dose of APVO436

Exclusion Criteria for Part 2: Dose Expansion Phase

Subjects with any of the following will not be eligible for study participation:

1. Acute promyelocytic leukemia (APL) with t(15;17) translocation
2. Absolute peripheral blood myeloblast count greater than 20,000/mm3 - may receive hydroxyurea to reduce and control the myeloblast count down prior to and during the first week of the first cycle of treatment with study drug if necessary if deemed medically necessary and appropriate by the treating physician
3. Patients with active central nervous system (CNS) involvement by AML will be excluded. A lumbar puncture does not need to be performed unless there is clinical suspicion of CNS involvement per investigator judgement. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS AML is allowed with the approval of the sponsor.
4. History of seizures
5. Prior anti-CD123 therapy with APVO436; prior anti-CD123 therapy with bispecific antibodies, recombinant fusion proteins or antibody-drug conjugates is allowed.
6. Prior allogeneic, unrelated or autologous hematopoietic stem cell transplantation is allowed only in Cohort 5. The transplant must have been performed more than 100 days before the date of dosing on this study without any Grade ≥2 graft-versus-host disease (GVHD) secondary to prior allogenic transplant. Patients must be > 100 days from transplant and have been on no immunosuppressive therapy for > 30 days. Topical corticosteroids for minor skin rash (<5% body surface area) is acceptable.
7. Prior allogeneic, unrelated or autologous hematopoietic stem cell transplantation is not allowed for Cohorts 1 to 4
8. Prior solid organ transplant is acceptable provided the patient is on no immunosuppressive therapy.
9. Any therapy or experimental treatment for AML within 7 days of the first dose of study drug. Must have recovered to Grade ≤ 1 from any Grade 2 to 4 toxicity from previous treatment. The use of hydroxyurea is acceptable and does not exclude the patient.
10. Active, uncontrolled infection requiring systemic therapy. If the infection is controlled or has resolved, maintenance and/or prophylactic systemic antimicrobials are permitted.
11. Major surgery within 3 weeks prior to first dose of study drug
12. Known to be positive for HIV, hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV)
13. Uncontrolled hypertension, defined as blood pressure ≥ 140/90 mm Hg despite maximum medical intervention
14. History of congenital long QT syndrome or torsades de pointes
15. Pathologic bradycardia or heart block (excluding first degree heart block)
16. Prolonged baseline QTc, defined as QTcF (Fredericia correction) interval >480 msec (including subjects with a bundle branch block)
17. History of ventricular arrhythmia (excluding PVCs)
18. Major surgery within 28 days prior to informed consent
19. Unstable angina pectoris within 28 days
20. Myocardial infarction and/or new ST elevation or depression or new Q wave on ECG within 6 months
21. Any history of stroke
22. Symptomatic congestive heart failure Class III or greater (New York Heart Association Functional Classification)
23. On full dose anti-coagulation defined as warfarin intended to raise the INR to 2-3
24. Major hemorrhagic event within 28 days requiring transfusion of packed red blood cells
25. Prior history of hypertensive crisis or hypertensive encephalopathy
26. Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture was performed to confirm the absence of leukemic blasts in the cerebrospinal fluid (CSF)
27. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
28. Any open wound
29. Pregnant and nursing subjects are excluded because the effects of APVO436 on a fetus or nursing child are unknown
30. Treatment with any anticancer therapy (standard or investigational) within the previous 14 days prior to the first dose of study drug. In addition, subjects must have fully recovered (NCI CTCAE Grade 1) from the clinically significant toxic effects of that treatment. The use of hydroxyurea in subjects with rapidly proliferating disease is allowed only during Cycle 1. Hydroxyurea is allowed prior to starting the study, and may be used for two weeks after dosing in Cycle 1 (e.g., Days 1-14 dosed with hydroxyurea)
31. Substance use disorder, psychiatric, cognitive, or any other condition that, in the opinion of the Investigator, would pose a risk to the patient's safety, may compromise the patient's ability to understand and comply with the protocol or provide informed consent, or interfere with the study evaluation, study participation, or follow-up
32. Any difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration, or may cause a safety concern for the patient
33. Any uncontrolled medical condition, including but not limited to:

    1. Uncontrolled hypertension
    2. Unstable angina
    3. Clinically significant arrhythmias not controlled by medication
    4. Uncontrolled metabolic disorders such as hypercalcemia
34. Any other active systemic malignancies. Exceptions: noninvasive non-melanoma skin cancer, in situ carcinoma, cervical intraepithelial neoplasia, and breast or prostate cancer that is well controlled with anti-hormonal therapy
35. Any current autoimmune disorder requiring immunosuppressive therapy with more than a replacement dose of corticosteroids (i.e., > 10 mg/day of prednisone or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Dose Escalation: Maximum Tolerated Dose | during first 28 to 35 days of treatment
  Identify the maximum tolerated dose in dose-escalation (Phase 1) by assessment of dose-limiting toxicities
Part 2 - Dose Expansion: Safety | during first 28 to 35 days of treatment
  The cumulative incidence of Grade 3-4 AEs, and SAEs, and the incidence of AES of interest (≥Grade 2 CRS, ≥Grade 2 Infusion related reaction, ≥2 cardiac toxicity and ≥2 neurotoxicity as complications of CRS) for safety

SECONDARY OUTCOMES:
Part 1 - Dose Escalation: Frequency and severity of adverse events as assessed by CTCAE v5.0 | Patient will be followed for the duration of treatment, an expected average of 6 months, and for up to 7 days following last treatment
  The safety profile of APVO436 will be assessed by monitoring incidence and severity of adverse events
Part 1 - Dose Escalation: Maximum serum drug concentration | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be obtained from all patients for determination of the maximum serum concentration of APVO436
Part 1 - Dose Escalation: Area under the concentration-time curve (AUC) | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be obtained from all patients for determination of the AUC of APVO436
Part 1 - Dose Escalation: Elimination of half-life | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be obtained from all patients for determination of the T1/2 of APVO436
Part 1 - Dose Escalation: Changes in T-cell populations to measure pharmacodynamics of APVO436 | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be collected from all patients and evaluated by flow cytometry for changes in T-cell populations
Part 1 - Dose Escalation: Changes in peripheral blasts to measure pharmacodynamics of APVO436 | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be collected from all patients and evaluated by flow cytometry for changes in peripheral blasts
Part 1 - Dose Escalation: Immunogenicity of APVO436 | Patient will have laboratory assessments prior to dosing on Day 1, throughout the study, and up to 7 days following last dose.
  Blood samples will be collected from all patients and tested for antibody formation to APVO436
Part 2 - Dose Expansion: Efficacy - Incidence of composite CR (CR + CRi + CRh) | Patient will have assessment at the end of each Cycle (each Cycle is 28 days) up to 2 years
  Incidence of composite CR (CR + CRi + CRh) in relapsed patients as a measure of efficacy within the confines of a Phase 1B study.
Part 2 - Dose Expansion: Efficacy - MRD Status | Patient will have assessment at the end of each Cycle (each Cycle is 28 days) up to 2 years
  Incidence of patients who are able to achieve MRD-negative CR
Part 2 - Dose Expansion: Efficacy - MRD Status | Patient will have assessment through study completion, an average of 1 year
  Incidence of patients who undergo HSCT post protocol therapy
Part 2 - Dose Expansion: Exploratory - LFS | Up to 2 years
  Leukemia-free survival (LFS)
Part 2 - Dose Expansion: Exploratory - 1-year LFS rate | 1 year
  1-year LFS rate;
Part 2 - Dose Expansion: Exploratory - 2-year LFS rate | 2 years
  2-year LFS rate;
Part 2 - Dose Expansion: Exploratory - MRD | 1 month and 4 months
  Pre- and Post-protocol therapy (after 1 cycle and after 4 cycles) MRD burden in Cohort 3 Percent Reduction of MRD in Cohorts 4 and 5 after 1 cycle and 4 cycles of protocol therapy

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - The University of Kansas Clinical Research Center, Westwood, Kansas
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Ohio State University Wexner Medical Center/James Cancer Hospital, Columbus, Ohio
  - Greenville Health System, Institute for Translational Oncology Research, Greenville, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Uckun FM, Lin TL, Mims AS, Patel P, Lee C, Shahidzadeh A, Shami PJ, Cull E, Cogle CR, Watts J. A Clinical Phase 1B Study of the CD3xCD123 Bispecific Antibody APVO436 in Patients with Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome. Cancers (Basel). 2021 Aug 15;13(16):4113. doi: 10.3390/cancers13164113. PMID 34439266
- [Result] Uckun FM, Watts J, Mims AS, Patel P, Wang E, Shami PJ, Cull E, Lee C, Cogle CR, Lin TL. Risk, Characteristics and Biomarkers of Cytokine Release Syndrome in Patients with Relapsed/Refractory AML or MDS Treated with CD3xCD123 Bispecific Antibody APVO436. Cancers (Basel). 2021 Oct 21;13(21):5287. doi: 10.3390/cancers13215287. PMID 34771451